CLINICAL TRIAL: NCT02413879
Title: An Evaluation of the Safety and Efficacy of the CleanCision Wound Retraction and Protection System in Protecting Surgical Incisions From Intraoperative Contamination When Used During Colorectal Surgery
Brief Title: Cleancision IntRaoperative Contamination prEvention Study
Acronym: CIRCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prescient Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLP-0001
Record Dates: First submitted 2015-03-27; First posted 2015-04-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Wound Contamination; Colorectal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): All study subjects will be treated using the CleanCision device.
  Interventions: Device: CleanCision

INTERVENTIONS:
Device: CleanCision — Wound protection during colorectal surgery.

SUMMARY:
This study entitled, An Evaluation of the Safety and Efficacy of the CleanCision Wound Retraction and Protection System in Protecting Surgical Incisions from Intraoperative Contamination When Used during Colorectal Surgery, is designed to evaluate contamination at the wound incision site when the CleanCision is used during surgery.

DETAILED DESCRIPTION:
This study entitled, An Evaluation of the Safety and Efficacy of the CleanCision Wound Retraction and Protection System in Protecting Surgical Incisions from Intraoperative Contamination When Used during Colorectal Surgery, is designed to evaluate bacterial contamination at the wound incision site when the CleanCision is used during surgery. The CleanCision is a surgical tool that is designed to be used for the primary purpose of protecting the wound from contamination that occurs to the incision site during surgery ultimately reducing the occurrence of Surgical Site Infections (SSI).

This is a prospective, multi-center, single-arm (non-randomized) clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* BMI 15-45, inclusive
* Colorectal surgery patient, planned resection
* Incision length meets labeling requirements
* Written informed consent using the governing IRB approved form

Exclusion Criteria:

* Patients with a pre-existing stoma
* Patients undergoing emergent colorectal surgery
* Known history of contact hypersensitivity or allergy to device materials
* Prior laparotomy or abdominal surgery within a timeframe that may present a safety risk or compromise study results
* Active infection, sepsis or systemic antibiotic therapy within timeframe that may impact safety or study results
* Active participation in any other clinical study of an experimental drug or device that may impact safety or study results
* Postsurgical life expectancy is less than the study follow up period
* Subject is pregnant or lactating
* Subject is under incarceration
* Subject considered to be inoperable following exploratory surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Papaconstantinou, MD, Principal Investigator — Scott & White Memorial Hospital
Locations (7):
- United States (7):
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Washington University Medical Center, St Louis, Missouri
  - Stony Brook Medicine, Stony Brook, New York
  - Baylor University Medical Center, Dallas, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Intermountain Healthcare McKay-Dee Hospital, Ogden, Utah

REFERENCES:
- [Derived] Papaconstantinou HT, Ricciardi R, Margolin DA, Bergamaschi R, Moesinger RC, Lichliter WE, Birnbaum EH. A Novel Wound Retractor Combining Continuous Irrigation and Barrier Protection Reduces Incisional Contamination in Colorectal Surgery. World J Surg. 2018 Sep;42(9):3000-3007. doi: 10.1007/s00268-018-4568-z. PMID 29523908

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 11 subjects in an initial study phase conducted at a single-center. The protocol was modified following this phase. Also, 11 subjects were in a pre-specified roll-in phase. The 22 participants in the Initial Study Phase and Roll-In Phase account for the discrepancy between Protocol Enrollment and Participant Flow "Started" value.
Groups:
- Treatment Group: All study subjects were treated using the CleanCision device.
Period: Overall Study
Arm/Group | Treatment Group
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: All study subjects will be treated using the CleanCision device.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 4
  White | 81
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 86
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.0 (5.8)
Medical History [Count of Participants; unit: Participants]
  IBD | 14
  Colorectal Cancer | 33
  Hypertension | 46
  Diabetes | 19
  History of Smoking | 46
  Steroid or other immunosuppressant within 1 month | 30

OUTCOME MEASURES:

1. Primary Outcome: Efficacy (Enteric Bacterial Contamination on the Exposed Surface of the CleanCision Sheath Compared to the Protected Incision Edge)
Description: Comparison of enteric bacterial contamination on the exposed surface of the CleanCision sheath compared to the protected incision edge
Time Frame: 1 day (end of the procedure and removal of the investigational device)
Population: Two subjects did not have swab results and thus were not included in the intention-to-treat analysis.
Measure: Number; unit: % of participants with contamination
Arm/Group | Treatment Arm
Number analyzed (Participants) | 84
% of participants with contamination
  Contamination Rate on Exposed Surface | 33.3
  Contamination Rate on Protected Incision Edge | 9.5
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority; p < 0.001, McNemar

2. Primary Outcome: Safety (Serious Adverse Events Directly Attributable to the Device)
Description: Incidence of Serious Adverse Events directly attributable to the device
Time Frame: 30 days
Population: All subjects within the Treatment arm were analyzed (Intention-to-treat).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 86
Participants | 0

3. Secondary Outcome: Efficacy (Bacterial Contamination on the Exposed Surface of the CleanCision Sheath Compared to the Protected Incision Edge)
Description: Comparison of bacterial contamination on the exposed surface of the CleanCision sheath compared to the protected incision edge
Time Frame: 1 day (end of the procedure and removal of the investigational device)
Population: Two subjects did not have swab results and thus were not included in the intention-to-treat analysis.
Measure: Number; unit: % of participants with contamination
Arm/Group | Treatment Arm
Number analyzed (Participants) | 84
% of participants with contamination
  Contamination Rate on Exposed Surface | 34.5
  Contamination Rate on Protected Incision Edge | 11.9
Statistical Analysis 1: Comparison: Treatment Arm; Test type: Superiority; p < 0.001, McNemar

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 17/86
Other Adverse Events (participants affected / at risk) | 10/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=86)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Infection (Infections and infestations) | 2 (2)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Intra-abdominal haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=86)
Vomiting (Gastrointestinal disorders) | 5 (5)
Urinary tract infection (Infections and infestations) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days